CLINICAL TRIAL: NCT02876159
Title: The Immunologic Basis for an Attenuated Immune Response to the Influenza Vaccine After Repeated Annual Vaccination
Acronym: FLU1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Mark Mulligan, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00090196
Record Dates: First submitted 2016-08-04; First posted 2016-08-23 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Influenza
Keywords: Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccination Naïve (Experimental): Participants who have received an influenza vaccine in 2 or less of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  Interventions: Biological: 2016-2017 Influenza Vaccine
- Vaccination Experienced (Experimental): Participants who have received an influenza vaccine at least 3 of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  Interventions: Biological: 2016-2017 Influenza Vaccine

INTERVENTIONS:
Biological: 2016-2017 Influenza Vaccine — Quadrivalent influenza A/Hemagglutinin Type 1 (H1N1), A/Influenza A virus subtype (A/H3N2) H3N2,and B virus vaccine for Intramuscular (IM) use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.

SUMMARY:
This is a prospective pilot study designed to suggest differences in the immunologic response to the seasonal influenza vaccine in people with regular vaccination history compared to those vaccinated less regularly. Participants will receive one dose of the Food and Drug Administration (FDA) approved 2016-2017 seasonal influenza vaccine. Immune system data will be collected at standard time points. The duration of the study for each participant will be approximately 1 month.

DETAILED DESCRIPTION:
This is a prospective pilot study in 20 males and non-pregnant females, 20 to 30 years old, inclusive, who are in good health and meet all eligibility criteria. The study is designed to evaluate differences in the immunologic response to the seasonal influenza vaccine in people with regular vaccination history compared to those vaccinated less regularly.

Participants will be sorted to either Arm A (Naïve) or Arm B (Experienced) based on their vaccination history. Those vaccinated no more than 2 out of the past 5 years will be in Arm A. Those vaccinated 3 or more out of the past 5 years will be in Arm B. Participants will receive one dose of the Food and Drug Administration (FDA) approved 2016-2017 seasonal influenza vaccine. The duration of the study for each participant will be approximately 1 month. Subjects will return for clinic visits on Days 3, 8, 15, and 29 during the month follow-up period following vaccination.

The study has two primary objectives; to evaluate the antibody response to the influenza vaccine in people who are vaccinated regularly and those vaccinated less regularly; the second is to evaluate circulating follicular helper T cells (TFH) in people who are vaccinated regularly and those vaccinated less regularly.

ELIGIBILITY:
Inclusion Criteria:

* Capable of informed consent and provision of written informed consent before any study procedures.
* Capable of attending all study visits according to the study schedule.
* Are in good health, as determined by medical history and targeted physical exam related to this history.
* Oral temperature is less than 38 degrees Celsius.
* Resting pulse rate is between 50 and 115 beats per minute.
* Female subjects of childbearing age must have a negative urine pregnancy test within 24 hours before study vaccination.
* Have received the influenza vaccine at least 3 of the past 5 years or have received the influenza vaccine in 2 or less of the past 5 years.

Exclusion Criteria:

* Have an acute illness within 72 hours before vaccination.
* Have any condition that, in the opinion of the principal investigator, would place the subject at an unacceptable risk of injury or confound the interpretation of the study results.
* Have any acute or chronic medical condition that, in the opinion of the principal investigator, would make vaccination unsafe or interfere with the evaluation of immune response to study vaccination.
* Have a suppressed immune system as a result of illness, immunosuppressive medication, chemotherapy, or radiation therapy within 3 years prior to study vaccination.
* Have known HIV, hepatitis B, or hepatitis C infection.
* Have a known history of autoimmune disease.
* Have taken oral or parenteral corticosteroids of any dose within 30 days before study vaccination.
* Have taken high-dose inhaled corticosteroids within 30 days before study vaccination.
* Have received any licensed live vaccine within 30 days or any licensed inactivated vaccine within 14 days prior to study vaccination.
* Have planned vaccination with any vaccine during the 29-day duration of subject study participation.
* Have received immunoglobulin or other blood products, with the exception of Rho D immunoglobulin, within 90 days prior to study vaccination.
* Have donated blood or blood products within 30 days before study vaccination, plan to donate blood at any time during the 29-day duration of subject study participation, or plan to donate blood within 30 days after the last blood draw.
* Have known hypersensitivity or allergy to eggs, egg protein, chicken protein, or other compounds of the study vaccine.
* Have a history of severe reactions following vaccination with influenza virus vaccines

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mulligan, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of the Emory Vaccine Center, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this study were enrolled from 07/01/2016 to 09/30/2016. Clinical study was conducted at Hope Clinic of Emory University.
Groups:
- Vaccination Naïve: Participants who have received an influenza vaccine in 2 or less of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  2016-2017 Influenza Vaccine: Quadrivalent influenza A/H1N1, A/H3N2, B virus vaccine for intramuscular use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.
- Vaccination Experienced: Participants who have received an influenza vaccine at least 3 of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  2016-2017 Influenza Vaccine: Quadrivalent influenza A/H1N1, A/H3N2, B virus vaccine for intramuscular use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.
Period: Overall Study
Arm/Group | Vaccination Naïve | Vaccination Experienced
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccination Naïve | Vaccination Experienced | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (1.9) | 24.6 (2.2) | 24.0 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 5 | 9 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.7 (8) | 22.8 (2.77) | 24.3 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Geometric Mean Serum Hemagglutination Inhibition (HAI) Antibody Titer
Description: Geometric mean serum HAI antibody titers serum HAI titer will be collected via blood draw. Titer for serum HAI antibodies will be calculated using the geometric mean. Change is defined as the difference in means from Day 1 to Day 29.
Time Frame: Baseline (Day 1), Day 29
Measure: Mean (Standard Deviation); unit: HAI antibody Titers
Groups:
- Vaccination Naïve: Participants who have received an influenza vaccine in 2 or less of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  2016-2017 Influenza Vaccine: Quadrivalent influenza A/Hemagglutinin Type 1 (H1N1), A/Influenza A virus subtype (H3N2), B virus vaccine for intramuscular use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.
- Vaccination Experienced: Participants who have received an influenza vaccine at least 3 of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  2016-2017 Influenza Vaccine: Quadrivalent influenza A/Hemagglutinin Type 1 (H1N1)/ Influenza A virus subtype H3N2, B virus vaccine for intramuscular use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.
Arm/Group | Vaccination Naïve | Vaccination Experienced
Number analyzed (Participants) | 10 | 10
HAI antibody Titers
  Day 1 | 23 (19.9) | 56.5 (95.7)
  Day 29 | 188 (191.4) | 108 (89)

2. Primary Outcome: Change in Mean Level of Circulating Follicular Helper T (TFH) Cells
Description: TFH cells will be collected via blood draw. Change is defined as the difference in the mean levels of cells from baseline, day 8, and day 15.
Time Frame: Up to 15 Days
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Vaccination Naïve | Vaccination Experienced
Number analyzed (Participants) | 10 | 10
cells/mm^3
  Day 1 | 1.9 (1) | 1.4 (0.8)
  Day 8 | 13.8 (11.4) | 2.96 (1.8)
  Day 15 | 4.1 (2.3) | 2.5 (4.1)

3. Secondary Outcome: Change in Mean Levels of Plasmablasts
Description: Plasmablasts will be collected via blood draw. Change is defined as the difference in mean levels from baseline to Day 29.
Time Frame: Up to 29 Days
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Vaccination Naïve | Vaccination Experienced
Number analyzed (Participants) | 10 | 10
cells/mm^3
  Day 1 | 2.5 (2.3) | 0.9 (0.7)
  Day 8 | 6.7 (5.1) | 0.5 (0.3)
  Day 15 | 2.3 (3.0) | 0.6 (0.3)

4. Secondary Outcome: Change in Mean Levels of Memory B Cells From Baseline (Day 1) to Day 29
Description: Memory B cells will be collected via blood draw. Change is defined as the difference in mean levels from baseline to Day 29.
Time Frame: Baseline (Day 1) and Day 29
Population: only 9 participant samples were analyzed as 1 sample could not be analyzed
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Vaccination Naïve | Vaccination Experienced
Number analyzed (Participants) | 9 | 9
cells/mm^3
  Day 1 | 0.18 (0.22) | 0.46 (0.72)
  Day 29 | 0.71 (0.77) | 0.29 (0.48)

5. Secondary Outcome: Change in Mean Levels of Antigen-specific IL-2 Producing CD4+ T Cells
Description: Antigen-specific Interleukin 2 (IL-2) producing cluster of differentiation 4 (CD4)+ T cells will be collected via blood draw. Change is defined as the difference in mean levels from baseline to Day 29.
Time Frame: Up to 29 Days
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- Vaccination Naive: Participants who have received an influenza vaccine in 2 or less of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  2016-2017 Influenza Vaccine: Quadrivalent influenza A/H1N1, A/H3N2, B virus vaccine for intramuscular use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.
Arm/Group | Vaccination Naive | Vaccination Experienced
Number analyzed (Participants) | 10 | 10
cells/mm^3
  Day 1 | 0.018 (0.02) | 0.018 (0.017)
  Day 29 | 0.013 (0.097) | 0.038 (0.024)

6. Secondary Outcome: Change in Mean Levels of Antigen-specific Cluster of Differentiation 8 (CD8) + T Cells
Description: CD8+T cells will be collected via blood draw. Change is defined as the difference in mean levels from baseline to Day 29.
Time Frame: Up to 29 Days
Population: CD8+T cell assays were not collected since the split virus influenza vaccine was not likely to induce any detectable CD8+ T cell responses.
Arm/Group | Vaccination Naive | Vaccination Experienced
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AE's) data was collected from the participant signing the informed consent to Day 29 post vaccination.
Groups:
- Vaccination Naïve: Participants who have received an influenza vaccine in 2 or less of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  2016-2017 Influenza Vaccine: Quadrivalent influenza A/H1N1, A/H3N2, B, B virus vaccine for intramuscular use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.
- Vaccination Experienced: Participants who have received an influenza vaccine at least 3 of the past 5 years will receive the FDA-approved 2016-2017 influenza vaccine.
  2016-2017 Influenza Vaccine: Quadrivalent influenza A/H1N1, A/H3N2, B, B virus vaccine for intramuscular use is a sterile, clear and slightly opalescent suspension administered as a single 0.5 mL intramuscular dose.
Arm/Group | Vaccination Naïve | Vaccination Experienced
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The numbers of subjects in this pilot study are small. A larger study will be required for confirmation of the outcome measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes